CLINICAL TRIAL: NCT03807804
Title: An Open-label, Standard Therapy as a Controlled, Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of HLCM051(MultiStem) in Patients With Acute Respiratory Distress Syndrome (ARDS) Caused by Pneumonitis
Brief Title: Efficacy and Safety Study of HLCM051(MultiStem®) for Pneumonic Acute Respiratory Distress Syndrome
Acronym: ONE-BRIDGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B04-02
Record Dates: First submitted 2019-01-08; First posted 2019-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: 【ARDS caused by pneumonia cohort】Parallel Assignment 【ARDS caused by COVID-19 cohort】Single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLCM051 group【ARDS caused by pneumonia cohort】 (Experimental): * Patients will receive the standard therapy
  * A single, one-time dose of HLCM051 9.0×108 (±20%) cells are intravenously infused as a naturally dropped single dose over 30 to 60 minutes at the maximum infusion speed of 10 mL/minute
  Interventions: Biological: HLCM051
- Standard treatment group【ARDS caused by pneumonia cohort】 (No Intervention): •Patients will receive the standard therapy
- HLCM051 group【ARDS caused by COVID-19 cohort 】 (Experimental): * Patients will receive the standard therapy
  * A single, one-time dose of HLCM051 9.0×108 (±20%) cells are intravenously infused as a naturally dropped single dose over 30 to 60 minutes at the maximum infusion speed of 10 mL/minute
  Interventions: Biological: HLCM051

INTERVENTIONS:
Biological: HLCM051 — HLCM051 is the stem cell product that can be mass-produced, being derived from adult adhesive stem cells that were taken from bone marrow of healthy unrelated donors from whom the informed consent was obtained, and proliferated ex vivo.
  Arms: HLCM051 group【ARDS caused by COVID-19 cohort 】; HLCM051 group【ARDS caused by pneumonia cohort】

SUMMARY:
The primary object of this clinical study is to investigate the efficacy of HLCM051 in patients with ARDS caused by pneumonitis.

DETAILED DESCRIPTION:
The objectives of this clinical study are as follows(ARDS caused by pneumonia cohort):

1. Primary objective To investigate the efficacy of HLCM051 in patients with ARDS caused by pneumonia
2. Secondary objective To confirm the safety of HLCM05 in patients with ARDS caused by pneumonia
3. Exploratory objective To investigate changes of biomarkers in patients with ARDS caused by pneumonia

The number of patients enrolled is 30 (20 patient in the HLCM051 group and 10 patients in the standard therapy group)

The objectives of this clinical study is as follows(ARDS caused by COVID-19 cohort):

1. Exploratory objective To investigate the safety and the efficacy of HLCM051 in patients with ARDS caused by SARS-Cov-2 infection

The number of patients enrolled is Approximately 5 (the HLCM051 group only)

ELIGIBILITY:
Inclusion Criteria(ARDS caused by pneumonia cohort):

1. Provision of informed consent by the patient or his/her legal representative in case the patient is incapable of giving consent due to sedation etc
2. Male or female aged 20 to 90 years at informed consent (Asians only)
3. Patients with ARDS caused by pneumonia of those who were diagnosed as having ARDS according to the Berlin Definition
4. Patients who are confirmed to have the following findings in the Berlin Definition within the same 24 hours 1)PaO2/FiO2 (P/F) ratio ≤ 300 mmHg with positive end-expiratory pressure (PEEP) ≥ 5 cmH2O 2)Bilateral opacities on chest X-ray or CT (not fully explained by effusions, lobar/lung collapse, and nodular shadow) 3)Respiratory failure that cannot be explained by cardiac failure and fluid overload
5. Patients who underwent chest high-resolution computed tomography (HRCT)
6. Patients with HRCT score ≥211 according to the abbreviated HRCT scoring system
7. Patients with APACHE II score <27 at the diagnosis of ARDS
8. Patients who underwent artificial respiration with intubation
9. Patients who can start receiving the investigational product within 72 hours (3 days) after the diagnosis of ARDS
10. Patients whose condition is expected to be stable for at least 4 hours after initiating investigational product administration "Stable" means the condition where there is no need for significant sustained increase in FiO2 or PEEP and the supportive care for the cardiovascular system is not required (e.g. an increase in the dose of norepinephrine or epinephrine by ≥0.1 mcg/kg/min or an increase in the dose of inotropic agent or vasopressor by ≥20% besides norepinephrine and epinephrine for blood pressure control)
11. Women who are neither pregnant, breastfeeding, planning to become pregnant during the study period. Women of childbearing potential must agree on the use of appropriate contraceptive methods under the guidance of investigators through the completion of the clinical study
12. Male patients who have female partners of childbearing potential must agree on the use of appropriate contraceptive methods under the guidance of investigators through the completion of the clinical study

Exclusion Criteria(ARDS caused by pneumonia cohort):

1. Patients without life expectancy of 48 hours
2. Patients who are under artificial dialysis at screening
3. Patients whose life expectancy is <6 months because of complications at screening
4. Patients under ventilator at home due to chronic respiratory disease
5. Patients who have been on mechanical ventilation for ≥ 1 week
6. Patients with obvious honeycomb lung at screening consistent with pre-existing late-stage interstitial lung disease
7. Patients with clinically evident findings consistent with diffuse alveolar hemorrhage
8. Patients with chronic respiratory disease that requires continuous domiciliary oxygen therapy
9. Patients with severe COPD (stage III or severe according to the GOLD Classification)
10. Patients with chronic pulmonary hypertension (class III or IV according to the World Health Organization Classification of Functional Status of Patients With Pulmonary Hypertension)
11. Patients with a history of lung lobectomy, single-lung pneumonectomy or pulmonary transplantation
12. Patients who are appropriate to be treated with extracorporeal membrane oxygenation (ECMO) at screening
13. Patients who were resuscitated after cardio-respiratory arrest
14. Patients with a history of ST-segment elevation myocardial infarction within 6 months before informed consent
15. Patients with mean arterial (blood) pressure (MAP) <60 mmHg despite treatment with one or more vasopressor or cardiotonic agent
16. Patients with severe chronic liver disease (Child-Pugh >10)
17. Patients with a history of transplantation with autologous or allogeneic, bone marrow or peripheral stem cells for other purposes than the treatment of hematological tumor
18. Patients with malignancy requiring treatment at screening
19. Patients infected with human immunodeficiency virus (HIV)
20. Patients with a history of acute allergic reaction to the preparations derived from human tissues, bovine or swine materials, and those who refuse the use of biological products due to religious reasons
21. Patients for whom ARDS is not judged as the chief complaint by the investigator (sub-investigator) based on clinical findings
22. Patients who received other investigational drugs or products within 30 days prior to informed consent
23. Patients who are participating or planned to participate in other clinical studies (except for observational clinical researches that do not require intervention) during this clinical study
24. Patients who are inappropriate to participate in this clinical study because of significant complications (such as pneumothorax ) or psychiatric disorders as judged by the investigator
25. Patients who is suspected SARS-CoV-2 infection

Inclusion Criteria(ARDS caused by COVID-19 cohort ):

1. Provision of informed consent by the patient or his/her legal representative in case the patient is incapable of giving consent due to sedation etc.
2. Male or female aged 20 to 70 years at informed consent (Asians only)
3. Patients tested positive for COVID-19
4. Patients with ARDS caused by COVID-19 of those who were diagnosed as having ARDS according to the Berlin Definition
5. Patients who are confirmed to have the following findings in the Berlin Definition within the same 24 hours 1)PaO2/FiO2 (P/F) ratio ≤ 300 mmHg with positive end-expiratory pressure (PEEP) ≥ 5 cmH2O 2)Bilateral opacities on chest X-ray or CT (not fully explained by effusions, lobar/lung collapse, and nodular shadow) 3)Respiratory failure that cannot be explained by cardiac failure and fluid overload
6. Patients who underwent Chest X-ray, chest CT or high-resolution computed tomography (HRCT) as far as possible
7. Patients with APACHE II score <27 at the diagnosis of ARDS
8. Patients who underwent artificial respiration with intubation
9. Patients who can start receiving the investigational product within 72 hours (3 days) after the diagnosis of ARDS
10. Women who are neither pregnant, breastfeeding, planning to become pregnant during the study period. Women of childbearing potential must agree on the use of appropriate contraceptive methods under the guidance of investigators through the completion of the clinical study
11. Male patients who have female partners of childbearing potential must agree on the use of appropriate contraceptive methods under the guidance of investigators through the completion of the clinical study

Exclusion Criteria(ARDS caused by COVID-19 cohort ):

1. Patients without life expectancy of 48 hours
2. Patients who are under artificial dialysis at screening
3. Patients whose life expectancy is <6 months because of complications at screening
4. Patients under ventilator at home due to chronic respiratory disease
5. Patients who have been on mechanical ventilation for ≥ 1 week
6. Patients with obvious honeycomb lung at screening consistent with pre-existing late-stage interstitial lung disease
7. Patients with clinically evident findings consistent with diffuse alveolar hemorrhage
8. Patients with chronic respiratory disease that requires continuous domiciliary oxygen therapy
9. Patients with severe COPD (stage III or severe according to the GOLD Classification)
10. Patients with chronic pulmonary hypertension (class III or IV according to the World Health Organization Classification of Functional Status of Patients With Pulmonary Hypertension)
11. Patients with a history of lung lobectomy, single-lung pneumonectomy or pulmonary transplantation
12. Patients who are appropriate to be treated with extracorporeal membrane oxygenation (ECMO) at screening
13. Patients who were resuscitated after cardio-respiratory arrest
14. Patients with a history of ST-segment elevation myocardial infarction within 6 months before informed consent
15. Patients with mean arterial (blood) pressure (MAP) <60 mmHg despite treatment with one or more vasopressor or cardiotonic agent
16. Patients with severe chronic liver disease (Child-Pugh >10)
17. Patients with a history of transplantation with autologous or allogeneic, bone marrow or peripheral stem cells for other purposes than the treatment of hematological tumor
18. Patients with malignancy requiring treatment at screening
19. Patients infected with human immunodeficiency virus (HIV)
20. Patients with a history of acute allergic reaction to the preparations derived from human tissues, bovine or swine materials, and those who refuse the use of biological products due to religious reasons
21. Patients for whom ARDS is not judged as the chief complaint by the investigator (sub-investigator) based on clinical findings
22. Patients who have used other investigational drugs or products within 30 days before informed consent (excluding other investigational drugs or products used for the purpose of treating COVID-19)
23. Patients who are participating or planning to participate in other clinical studies during the study period (excluding other clinical studies, clinical researches and observational clinical researches that do not require intervention for the purpose of treating COVID-19)
24. Patients who are inappropriate to participate in this clinical study because of significant complications (such as pneumothorax ) or psychiatric disorders as judged by the investigator

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days (VFD)(ARDS caused by pneumonia cohort) | 28 days after administration of the investigational product
  VFD for 28 days after administration of the investigational product
Adverse events(ARDS caused by COVID-19 cohort) | From informed consent to 180 days after administration of the investigational product
  The number and rate of adverse events
Change from baseline in systolic blood pressure(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in systolic blood pressure(mmHg)
Change from baseline in diastolic blood pressure(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in diastolic blood pressure(mmHg)
Change from baseline in pulse rate(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in pulse rate(beats/min)
Change from baseline in respiration(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in respiration(breath/min)
Change from baseline in oxygen saturation(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in oxygen saturation(%)
Change from baseline in body temperature(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in body temperature(C)
Change from baseline in red blood cell count(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in red blood cell count(/uL)
Change from baseline in hemoglobin(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in hemoglobin(g/dL)
Change from baseline in hematocrit(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in hematocrit(%)
Change from baseline in leukocyte count(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in leukocyte count(/uL)
Change from baseline in neutrophils(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in neutrophils(%)
Change from baseline in eosinophils(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in eosinophils(%)
Change from baseline in basophils(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in basophils(%)
Change from baseline in lymphocytes(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in lymphocytes(%)
Change from baseline in monocytes(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in monocytes(%)
Change from baseline in platelet count(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in platelet count(/uL)
Change from baseline in asparate aminotransferase(AST)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in asparate aminotransferase(AST)(IU/L)
Change from baseline in alanine aminotransferase(ALT)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in alanine aminotransferase(ALT)(IU/L)
Change from baseline in alkaline phosphatase(ALP)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in alkaline phosphatase(ALP)(IU/L)
Change from baseline in total bilirubin(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in total bilirubin(mg/dL)
Change from baseline in blood urea nitrogen(BUN)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in blood urea nitrogen(BUN)(mg/dL)
Change from baseline in creatinine(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in creatinine(mg/dL)
Change from baseline in sodium(Na)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in sodium(Na)(mmol/L)
Change from baseline in potassium(K)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in potassium(K)(mmol/L)
Change from baseline in chloride(Cl)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in chloride(Cl)(mmol/L)
Change from baseline in calcium(Ca)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in calcium(Ca)(mg/dL)
Change from baseline in blood sugar(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in blood sugar(mg/dL)
Change from baseline in urinary protein(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in urinary protein(- to >= 4+)
Change from baseline in urinary sugar(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in urinary sugar(- to >= 4+)
Change from baseline in uric blood(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in uric blood(- to >= 4+)
Change from baseline in urinary sediment(RBC)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in urinary sediment(RBC)(/HPF)
Change from baseline in urinary sediment(WBC)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in urinary sediment(WBC)(/HPF)
Change from baseline in urinary sediment(Other)(ARDS caused by COVID-19 cohort) | From screening to 180 days after administration of the investigational product
  Change from baseline in urinary sediment(Other)(/HPF)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuya Ichikado, M.D., Ph.D., Principal Investigator — Saiseikai Kumamoto Hospital; Satoru Hashimoto, M.D., Ph.D., Principal Investigator — University Hospital, Kyoto Prefectural University of Medicine
Locations (29):
- Japan (29):
  - Investigational Site Number 027, Nagoya, Aichi-ken
  - Investigational Site Number 028, Nagoya, Aichi-ken
  - Investigational Site Number 005, Seto, Aichi-ken
  - Investigational Site Number 020, Toyoake, Aichi-ken
  - Investigational Site Number 003, Hirosaki, Aomori
  - Investigational Site Number 007, Iizuka, Fukuoka
  - Investigational Site Number 019, Ōgaki, Gifu
  - Investigational Site Number 011, Sapporo, Hokkaido
  - Investigational Site Number 010, Kobe, Hyōgo
  - Investigational Site Number 013, Kobe, Hyōgo
  - Investigational Site Number 017, Takarazuka, Hyōgo
  - Investigational Site Number 025, Yokohama, Kanagawa
  - Investigational Site Number 029, Yokohama, Kanagawa
  - Investigational Site Number 018, Kashihara, Nara
  - Investigational Site Number 026, Suita, Osaka
  - Investigational Site Number 022, Ōtsu, Shiga
  - Investigational Site Number 014, Izumo, Shimane
  - Investigational Site Number 024, Bunkyō-Ku, Tokyo
  - Investigational Site Number 021, Chuo Ku, Tokyo
  - Investigational Site Number 009, Itabashi-ku, Tokyo
  - Investigational Site Number 006, Minato-Ku, Tokyo
  - Investigational Site Number 004, Shinagawa-Ku, Tokyo
  - Investigational Site Number 008, Shinjuku-Ku, Tokyo
  - Investigational Site Number 023, Shinjuku-Ku, Tokyo
  - Investigational Site Number 012, Hiroshima
  - Investigational Site Number 001, Kumamoto
  - Investigational Site Number 002, Kyoto
  - Investigational Site Number 015, Nagasaki
  - Investigational Site Number 016, Saga

REFERENCES:
- [Derived] Ichikado K, Kotani T, Kondoh Y, Imanaka H, Johkoh T, Fujimoto K, Nunomiya S, Kawayama T, Sawada M, Jenkins E, Tasaka S, Hashimoto S. Clinical efficacy and safety of multipotent adult progenitor cells (invimestrocel) for acute respiratory distress syndrome (ARDS) caused by pneumonia: a randomized, open-label, standard therapy-controlled, phase 2 multicenter study (ONE-BRIDGE). Stem Cell Res Ther. 2023 Aug 22;14(1):217. doi: 10.1186/s13287-023-03451-z. PMID 37608287